CLINICAL TRIAL: NCT05963919
Title: Determinants of Functional Capacity in Children With Asthma
Status: Completed | Type: Observational
Sponsor: Atlas University (Other)
Responsible Party: Sponsor
Other Study IDs: Atlasumkaya01
Record Dates: First submitted 2023-07-18; First posted 2023-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Asthma in Children
MeSH Terms: interventions — Respiratory Physiological Phenomena

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Asthma Group: 6 minute walk test, Pulmonary function test, Respiratory muscle strength test, Lower extremity muscle strength test
  Interventions: Other: 6-minute walk test; Other: Pulmonary function test; Other: Respiratory muscle strength test; Other: Lower extremity muscle strength test
- Control Group: 6 minute walk test, Pulmonary function test, Respiratory muscle strength test, Lower extremity muscle strength test
  Interventions: Other: 6-minute walk test; Other: Pulmonary function test; Other: Respiratory muscle strength test; Other: Lower extremity muscle strength test

INTERVENTIONS:
Other: 6-minute walk test — Functional capacity will be assessed with the 6-minute walk test (6MWT). 6MWT will be performed in accordance with the criteria of the American Thoracic Society. The 6MWT distance will be recorded in meters.
Other: Pulmonary function test — Pulmonary function test will be performed with a spirometer ("COSMED Pony FX" (COSMED; Italy) by ATS/ERS criteria. Forced expiratory volume in 1 second (FEV1) and peak expiratory volume (PEF) parameters will be measured. The results will be recorded both as a percentage of measured values and expected values.
Other: Respiratory muscle strength test — Respiratory muscle strength will be measured in accordance with ATS/ERS criteria using an electronic, mobile, (MicroRPM, Micro Medical; UK) intraoral pressure measuring device. Maximal inspiratory pressure (MIP) and maximal expiratory pressure (MEP) values will be recorded. Three measurements will be repeated for each maneuver and the highest value recorded as cmH2O.
Other: Lower extremity muscle strength test — The 30-Second Chair Test is administered using a folding chair without arms, with a seat height of 17 inches (43.2 cm). The chair, with rubber tips on the legs, is placed against a wall to prevent it from moving. The participant is seated in the middle of the chair, back straight; feet approximately a shoulder width apart, and placed on the floor at an angle slightly back from the knees, with one foot slightly in front of the other to help maintain balance. Arms are crossed at the wrists and held against the chest. The participant is encouraged to complete as many full stands as possible within 30 seconds. The participant is instructed to fully sit between each stand.

SUMMARY:
The primary aim of this study is to compare the respiratory function, respiratory muscle strength, functional capacity, and lower extremity strength of children with asthma and healthy children in the same age group. The secondary aim of our study is to determine the determinants of functional capacity in children with asthma.

ELIGIBILITY:
Asthma Group Inclusion Criteria:

* Being between the ages of 6-17
* Being diagnosed with asthma
* Able to walk, cooperate and clinically stable
* Being a volunteer to participate in the study
* To be able to speak, read, understand, and cooperate in Turkish

Asthma Group Exclusion Criteria:

* History of previous lung or liver transplant
* Having an acute exacerbation and/or a history of hospitalization in the last 1 month
* Having diagnosed orthopedic problems affecting mobility or a history of musculoskeletal surgery

Control Group Inclusion Criteria:

* Being between the ages of 6-17
* To be able to speak, read, understand, and cooperate in Turkish
* Being a volunteer to participate in the study

Control Group Exclusion Criteria:

* Having a diagnosed vision, hearing, or neurological disease that may affect balance
* Having any other neurological, orthopedic, cardiovascular, thoracic, or metabolic disease or pathological condition that would affect assessments
* Resting saturation below 90% during exercise tests

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children with asthma aged between 6-17 years and healthy children aged between 6-17 years will be included in the study. Informed consent forms for the study prepared for both the asthma group and the control group will be carefully explained and the participants will be included in the study after they and their parents have read, understood, and accepted.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
6-minute walk test | 15-20 minutes
Forced expiratory volume in 1 second (FEV1) | 10-15 minutes
Peak expiratory flow (PEF) | 10-15 minutes
Maximal inspiratory pressure (MIP) | 15-20 minutes
Maximal expiratory pressure (MEP) | 15-20 minutes
Lower extremity muscle strength | 5-10 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Atlas University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No